CLINICAL TRIAL: NCT01575054
Title: BOTOX® Treatment in Adult Patients With Post-Stroke Lower Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-116; 2011-004980-63 (EudraCT Number)
Record Dates: First submitted 2012-04-09; First posted 2012-04-11 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-08

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- botulinum toxin Type A (Experimental): Double-Blind Study Phase (12 weeks): On Day 1, botulinum toxin Type A 300 U will be given by intramuscular injections into specified muscles of the lower limb, and an optional dose of 100 U may be injected into additional lower limb muscles. Open Label Study Phase: Up to 3 treatments with botulinum toxin Type A up to 400 U will be given by intramuscular injections to the lower limb approximately every 12 weeks over a 42 week period.
  Interventions: Biological: botulinum toxin Type A
- Normal Saline (Placebo) Followed by botulinum toxin Type A (Other): Double-Blind Study Phase (12 weeks): On Day 1, normal saline (placebo) will be given by intramuscular injections into specified muscles of the lower limb, and optional injections may be administered into additional lower limb muscles. Open Label Study Phase: Up to 3 treatments with botulinum toxin Type A up to 400 U will be given by intramuscular injections to the lower limb approximately every 12 weeks over a 42 week period.
  Interventions: Biological: botulinum toxin Type A; Drug: Normal Saline

INTERVENTIONS:
Biological: botulinum toxin Type A — Double-Blind Study Phase (12 weeks): On Day 1, botulinum toxin Type A 300 U will be given by intramuscular injections into specified muscles of the lower limb, and an optional dose of 100 U may be injected into additional lower limb muscles. Open Label Study Phase: Up to 3 treatments with botulinum toxin Type A up to 400 U will be given by intramuscular injections to the lower limb approximately every 12 weeks over a 42 week period.
  Other Names: BOTOX®; onabotulinumtoxin A
Drug: Normal Saline — Double-Blind Study Phase (12 weeks): On Day 1, normal saline (placebo) will be given by intramuscular injections into specified muscles of the lower limb, and optional injections may be administered into additional lower limb muscles.
  Arms: Normal Saline (Placebo) Followed by botulinum toxin Type A

SUMMARY:
This study will evaluate the safety and efficacy of BOTOX® in the treatment of adult post-stroke lower limb spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of post-stroke lower limb spasticity for at least 3 months
* Minimum body weight of 50 kg
* Never treated with botulinum toxin of any serotype for any reason, or if previously treated with botulinum toxin of any serotype, if previously treated for spasticity in the affected lower limb, must have been administered

  * 20 weeks before Day 1, or if previously treated for any other indication must have been administered ≥12 weeks prior to Day 1

Exclusion Criteria:

* Spasticity in the opposite leg that requires treatment
* Casting of the study limb within 6 months or planned casting during the first 12 weeks of the study
* Treatment modalities in the study limb including ultrasound, electrical nerve stimulation, electrical stimulation, acupuncture within 1 month of Day 1 or treatments planned during the study
* Not able to perform 10 meter walking test independently with or without assistive device
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2012-05; Primary Completion 2014-09 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (12):
- United States (2):
  - Downey, California
  - Daytona Beach, Florida
- Montreal, Quebec, Canada
- Prague, Czechia
- Germany (2):
  - Wiesbaden
  - Würzburg
- Budapest, Hungary
- Krakow, Poland
- Krasnoyarsk, Russia
- Gyeonggi-do, South Korea
- United Kingdom (2):
  - Stoke-on-Trent, England
  - Fazakerley, Liverpool

REFERENCES:
- [Derived] Wein T, Esquenazi A, Jost WH, Ward AB, Pan G, Dimitrova R. OnabotulinumtoxinA for the Treatment of Poststroke Distal Lower Limb Spasticity: A Randomized Trial. PM R. 2018 Jul;10(7):693-703. doi: 10.1016/j.pmrj.2017.12.006. Epub 2018 Jan 9. PMID 29330071

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A | Normal Saline (Placebo) Followed by Botulinum Toxin Type A
Started | 233 | 235
Completed | 204 | 209
Not Completed | 29 | 26
Not completed — Other Reasons | 5 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Personal Reasons | 10 | 11
Not completed — Lost to Follow-up | 3 | 3
Not completed — Adverse Event | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | Normal Saline (Placebo) Followed by Botulinum Toxin Type A | Total
Number analyzed (Participants) | 233 | 235 | 468
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (12.60) | 57.0 (11.88) | 56.5 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 80 | 165
  Male | 148 | 155 | 303

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Ashworth Scale-Bohannon (MAS-B) Score of Ankle Plantar Flexors Using a 6-Point Scale
Description: The MAS-B is a 6-point scale used to evaluate spasticity based on grading the resistance encountered in the ankle flexors by passively moving the ankle plantar flexor muscles through their range of motion. The score ranges from 0 (no increase in muscle tone) to 4 (affected part(s) rigid in flexion or extension). Scores are converted to a 0 to 5 grade. The average of the weeks 4 and 6 MAS-B ankle change from baseline is the primary end point. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, 6 Weeks
Population: Intent-to-Treat: all randomized patients who were analyzed according to randomization assignment, regardless of treatment actually received
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A | Normal Saline (Placebo) Followed by Botulinum Toxin Type A
Number analyzed (Participants) | 233 | 235
Scores on a Scale
  Baseline | 4.1 (0.27) | 4.1 (0.25)
  Change from Baseline at 6 weeks | -0.81 (0.874) | -0.61 (0.835)

2. Secondary Outcome: Clinical Global Impression (CGI) of Overall Change by Physician Using a 9-Point Scale
Description: The CGI is a 9-point scale evaluating change from baseline status by the Physician. Scores range from +4 (very marked improvement) to -4 (very marked worsening). The average of the weeks 4 and 6 CGI by Physician score is used as a secondary end point. Higher scores indicate a greater improvement from baseline.
Time Frame: Baseline, 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A | Normal Saline (Placebo) Followed by Botulinum Toxin Type A
Number analyzed (Participants) | 233 | 235
Scores on a Scale | 0.86 (0.953) | 0.65 (0.902)

3. Secondary Outcome: Goal Attainment Scores on the 6-Point Physician-Assessed Goal Attainment Scale (GAS)
Description: The physician-assessed GAS is an individualized, goal-oriented 6-point scale used to track functional improvement toward active and passive goals. GAS scoring ranged from -3 to 2 (-3 = worse than start; 0 = expected goal/attained the defined therapeutic goal; 2 = much more than expected/improvements clearly exceeded the defined therapeutic goal). Active and Passive Goal scores are presented.
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A | Normal Saline (Placebo) Followed by Botulinum Toxin Type A
Number analyzed (Participants) | 233 | 235
Scores on a Scale
  Active Goals (N=226, 228) | -0.8 (1.34) [-0.99 to -0.56] | -1.0 (1.33) [-1.19 to -0.76]
  Passive Goals--use (N=214, 217) | -0.5 (1.42) [-0.77 to -0.31] | -0.8 (1.33) [-1.01 to -0.57]

4. Secondary Outcome: Change From Baseline in Average Pain Score While Walking on the 11-Point Pain Scale
Description: The patient is asked to select a number that best describes his/her pain while walking on an 11-point scale from 0 = "no pain" to 10 = "pain as bad as can be imagined". Patients are instructed to recall their average pain in the study limb during the 48-hour period prior to the visit. Patients with a baseline pain score >0 are included in the analyses.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A | Normal Saline (Placebo) Followed by Botulinum Toxin Type A
Number analyzed (Participants) | 180 | 164
Scores on a Scale
  Baseline | 4.5 (1.95) | 4.5 (2.13)
  Change from Baseline at Week 6 (N=175, 158) | -0.8 (2.30) | -1.1 (2.38)

5. Secondary Outcome: Change From Baseline in Modified Ashworth Scale-Bohannon (MAS-B) Score of Optional Muscles Using a 6-Point Scale
Description: The MAS-B is a 6-point scale used to evaluate spasticity based on grading the resistance encountered in the optional muscles by passively moving the muscles through their range of motion. Optional muscles treated include: Rectus Femoris, Flexor Digitorum Longus, Flexor Hallucis Longus, and Extensor Hallucis. The scores range from 0 (no increase in muscle tone) to 4 (affected part(s) rigid in flexion or extension). Scores are converted to a 0 to 5 grade. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A | Normal Saline (Placebo) Followed by Botulinum Toxin Type A
Number analyzed (Participants) | 143 | 133
Scores on a Scale
  Baseline Rectus Femoris (N=25, 25) | 3.3 (0.58) | 3.2 (0.59)
  Chng from BL at Wk6 in Rectus Femoris (N=24,25) | -0.9 (0.87) | -1.0 (1.14)
  Baseline Flexor Digitorum Longus (N=86,88) | 3.3 (0.76) | 3.4 (0.70)
  Chng from BL at Wk6 in Digitorum Longus (N=85,84) | -0.9 (1.11) | -0.8 (1.22)
  Baseline Flexor Hallucis Longus (N=73,67) | 3.1 (0.81) | 3.2 (0.83)
  Chng frm BL at Wk6 Flexor Hallucis Longus(N=72,66) | -1.0 (1.30) | -0.6 (1.20)
  Baseline Extensor Hallucis (N=23,13) | 3.6 (0.49) | 3.6 (0.51)
  Chng from BL at Wk6 in Extensor Hallucis (N=23,13) | -1.3 (1.22) | -1.3 (1.09)

ADVERSE EVENTS:
Description: The safety population during the 12-week double-blind phase included all enrolled patients who received at least 1 treatment injection in the study. The double-blind safety population is used to assess adverse events and serious adverse events.
Groups:
- Botulinum Toxin Type A: Double-Blind Study Phase (12 weeks): On Day 1, botulinum toxin Type A 300 U will be given by intramuscular injections into specified muscles of the lower limb, and an optional dose of 100 U may be injected into additional lower limb muscles.
- Normal Saline (Placebo): Double-Blind Study Phase (12 weeks): On Day 1, normal saline (placebo) will be given by intramuscular injections into specified muscles of the lower limb, and optional injections may be administered into additional lower limb muscles.
Arm/Group | Botulinum Toxin Type A | Normal Saline (Placebo)
Serious Adverse Events (participants affected / at risk) | 10/231 | 9/233
Other Adverse Events (participants affected / at risk) | 0/231 | 0/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=231) | Normal Saline (Placebo) (N=233)
Bifascicular block (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Barbiturates positive (Investigations) | 1 | 0
Opiates positive (Investigations) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 0
Drug abuse (Psychiatric disorders) | 1 | 0
Schizoaffective disorder (Psychiatric disorders) | 1 | 0
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.